CLINICAL TRIAL: NCT05206201
Title: A Phase 1, Prospective, Randomized, Double Blind, Parallel, Placebo-Control, Study Of Zy-19489 Administered Via Oral Route To Investigate The Safety, Tolerability And Pharmacokinetics In Healthy Adult Human Subjects
Brief Title: A Study Of Zy-19489 Administered Via Oral Route To Investigate The Safety, Tolerability And Pharmacokinetics In Healthy Adult Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZY19489 1001
Record Dates: First submitted 2021-08-04; First posted 2022-01-25 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2021-07

CONDITIONS: Malaria
Keywords: Malaria
MeSH Terms: conditions — Malaria | interventions — ZY-19489

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZY19489 Capsule (Experimental): Experimental study drug
  Interventions: Drug: ZY19489 Capsule
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: ZY19489 Capsule — Two part study with single and multiple dose
  Arms: ZY19489 Capsule
Drug: Placebo Capsule — Two part study with single and multiple dose
  Arms: Placebo

SUMMARY:
A Randomized, Double Blind, Parallel, Placebo-Control, Study Of ZY-19489 Administered Via Oral Route To Investigate The Safety, Tolerability And Pharmacokinetics In Healthy Adult Human Subjects aged between 18-55 years old (Both Inclusive).

DETAILED DESCRIPTION:
Study will conduct in two parts. In Part 1; single cohort of 8 subjects. Subjects will be enrolled within a 28 day screening period to ensure subjects meet all the inclusion criteria and none of the exclusion criteria. Subjects will be randomized in a ratio of 6:2 to receive single dose of ZY-19489 or placebo orally after an overnight fast of at least 10 hours.

In Part 2: study each cohort containing eight subjects will be given either a ZY19489 capsule or placebo for three consecutive days. Total three cohorts are planned in this study. Dose escalation will be performed for subsequent cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (non-pregnant, non-lactating) aged 18 to 55 years inclusive who will be contactable and available for the duration of the trial and up to 2 weeks following the End of Study visit.
2. Total body weight greater than or equal to 50 kg, and a body mass index (BMI) within the range of 18.5 to 30.0 kg/m2 (Both inclusive). BMI is an estimate of body weight adjusted for height. It is calculated by dividing the weight in kilograms by the square of the height in meters.
3. Certified as healthy by a comprehensive clinical assessment (detailed medical history, complete physical examination and special investigations).
4. Screening vital signs:

   Systolic blood pressure (SBP) - 90-140 mmHg, Diastolic blood pressure (DBP) - 60-90 mmHg, Heart rate (HR) 60-90 bpm.
5. QTcF ≤450 ms, PR interval ≤220 ms.
6. Female subjects with history of sterility or at least 1 year menopause or use of long acting non hormonal contraceptive measures (e.g., intrauterine device) and be willing and able to continue contraception for 90 days after administration of study treatment.
7. Male subjects must agree to use adequate contraception methods during the study and be willing and able to continue contraception for 90 days after administration of study treatment.
8. Completion of the written informed consent process prior to undertaking any study related procedure.
9. Must be willing and able to communicate and participate in the whole study.

Exclusion Criteria:

1. Haematology, clinical chemistry or urinalysis results at screening that are outside of clinically acceptable laboratory ranges, and are considered clinically significant by the Investigator.
2. Participation in any investigational product study within the 12 weeks preceding IMP administration.
3. History or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies, or history of anaphylaxis or other severe allergic reactions. Subjects with seasonal allergies/hay fever or allergy to animals or house dust mite that are untreated and asymptomatic can be enrolled in the study based on Investigator's discretion.
4. History of convulsion (including intravenous drug or vaccine-induced episodes). A medical history of a single febrile convulsion during childhood is not an exclusion criterion.
5. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immuno-deficiencies), insulin-dependent and non-insulin dependent diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, porphyria, psoriasis, rheumatoid arthritis, asthma (excluding childhood asthma, or mild asthma with preventative asthma medication required less than monthly), epilepsy, or obsessive-compulsive disorder.
6. History of malignancy of any organ system treated or untreated, within 5 years of screening, regardless of whether there is evidence of local recurrence or metastases.
7. Subjects with history of schizophrenia, bi-polar disease, psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis.
8. Subjects who have received psychiatric medications within 1 year prior to enrolment, or who have been hospitalized within 5 years prior to enrolment for either a psychiatric illness or due to danger to self or others.
9. History of more than one previous episode of major depression, any previous single episode of major depression lasting for or requiring treatment for more than 6 months, or any episode of major depression during the 5 years preceding screening.
10. History of recurrent headache (e.g. tension-type, cluster or migraine) with a frequency of ≥2 episodes per month on average and/or severe enough to require medical therapy, during the 5 years preceding screening.
11. Presence of clinically significant infectious disease or fever (e.g. sublingual temperature ≥38.5°C) within the 14 days prior to enrollment.
12. Evidence of acute illness within the 4 weeks prior to screening that the Investigator deems may compromise subject safety.
13. Significant inter-current disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, gastrointestinal, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
14. Subject has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion (e.g. gastrectomy, diarrhoea).
15. Blood donation of any volume within 1 month before IMP administration, or participation in any research study involving blood sampling (more than 450 mL/unit of blood), or blood donation to blood bank during the 12 weeks prior to IMP administration.
16. Medical requirement for intravenous immunoglobulin or blood transfusions within 3 months prior to enrollment.
17. History or presence of alcohol abuse (alcohol consumption more than 40 g/4 units/4 standard drinks per day), or drug habituation, or any prior intravenous usage of an illicit substance in past one year.
18. Tobacco use of more than 5 cigarettes or equivalent per day since last one year, and unable to stop smoking for the duration of the clinical unit confinement.
19. Female subject who is breastfeeding or currently pregnant or found positive on pregnancy test.

    Interfering substances
20. Any vaccination within the last 28 days and planned vaccination till final study visit.
21. Any corticosteroids, anti-inflammatory drugs (excluding commonly used over-thecounter anti-inflammatory drugs such as ibuprofen, acetylsalicylic acid, diclofenac), immunomodulators or anticoagulants within the past 3 months. Any subject currently receiving or having previously received immunosuppressive therapy (including systemic steroids, adrenocorticotrophic hormone or inhaled steroids) at a dose or duration potentially associated with hypothalamic-pituitary-adrenal axis suppression within the past year.
22. Ingestion of any poppy seeds within the 24 hours prior to screening
23. Consumption of beverages or food containing xanthine bases including Red Bull, chocolate, coffee etc. from 48 hours prior to enrollment.
24. Unwillingness to abstain from consumption of grapefruit or Seville oranges from 7 days prior to enrollment until the end of study.
25. Use of prescription drugs (excluding contraceptives) or non-prescription drugs or herbal supplements (such as St John's Wort), within 14 days or 5 half-lives (whichever is longer) prior to IMP dosing. Limited use of other non-prescription medications or dietary supplements, not believed to affect subject safety or the overall results of the study, may be permitted on a case-by- case basis following approval by the Sponsor in consultation with the Investigator. Subjects are requested to refrain from taking non-approved concomitant medications from recruitment until the conclusion of the study.
26. Any subject who, in the judgment of the Investigator, is likely to be non-compliant during the study, or is unable to cooperate because of a language problem or poor mental development.
27. Any subject who is the Principal Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
28. Any subject without a good peripheral venous access.
29. Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
30. Positive urine drug test.
31. Positive urine alcohol/breath alcohol test.
32. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.

    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This includes subjects with any of the following (at screening):
    * Sinus node dysfunction.
    * Complete bundle branch block.
    * Abnormal T wave morphology.
    * Any other ECG abnormalities in the standard 12-lead ECG in the opinion of the Investigator will interfere with the ECG analysis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse event of ZY-19489 administered to healthy subjects. | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Common Terminology Criteria for Adverse Event (CTCAE) (Version 5.0 or higher) system will be used for reporting and grading

SECONDARY OUTCOMES:
Area under the curve from the time of dosing to the last measurable concentration (AUC0-t) | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
Cmax | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
To assess the effect of ZY-19489/ZY-20486on the QTc interval (concentration/QTc modelling). | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  • Difference between baseline corrected QTc following placebo and baseline corrected QTc following ZY-19489
AUC0-∞ | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
Tmax | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
T1/2 | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
CL/F | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
VZ/F | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
λ | For Part 1 : Baseline to Day 28 and For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
AUC0-24 | For Part 2 : Baseline to Day 30
  AUC0-24 after first dose on Day 0 will be calculated with PK samples on Day 01. AUC0-24 after third dose on Day 2 will be calculated with PK samples on Day 03
Accumulation Index | For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
Rac(AUC) | For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486
Rac(Cmax) | For Part 2 : Baseline to Day 30
  Estimation of ZY-19489 and its metabolite ZY-20486

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deven Parmar, MD, Study Chair — Zydus Therapeutics Inc.
Locations (1):
- Zydus Research Centre, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No